CLINICAL TRIAL: NCT07287709
Title: Evaluation Of Laser Versus Conventional Pulpotomies In Mature Molar Teeth With Irreversible Pulpitis (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation Of Laser Versus Conventional Pulpotomies In Mature Molar Teeth With Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rana Hegaz (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Rana Hegaz, Assistant lecturer ,Endodontics, Department of Conservative Dentistry, Faculty of Dentistry, Alexandria University, Alexandria, Egypt., Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9258137
Record Dates: First submitted 2025-11-23; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Irreversible Pulpitis (Toothache)
Keywords: Photobiomodulation,; photocoagulation,; pulpotomy,; segmentation,; irreversible pulpitis; artificial intelligence; bioceramic putty
MeSH Terms: conditions — Toothache | interventions — Lasers, Semiconductor; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A Photo-biomodulation pulpotomy with Bioceramic putty (Experimental)
  Interventions: Device: Diode laser
- Group B photocoagulation pulpotomy with Bioceramic putty (Experimental)
  Interventions: Device: Diode laser
- Group C(Control) Conventional pulpotomy with Bioceramic putty (Active Comparator)
  Interventions: Other: Sodium Hypochlorite Solution

INTERVENTIONS:
Device: Diode laser — a contact-type laser, it selectively and precisely affects only the tissues directly beneath it, thereby preserving the surrounding radicular tissue
  Arms: Group A Photo-biomodulation pulpotomy with Bioceramic putty; Group B photocoagulation pulpotomy with Bioceramic putty
Other: Sodium Hypochlorite Solution — A disinfecting agent used in conventional pulpotomy procedures
  Arms: Group C(Control) Conventional pulpotomy with Bioceramic putty

SUMMARY:
this clinical trial is evaluating the outcome of laser assisted pulpotomy compared to conventional pulpotomy in mature teeth with symptomatic irreversible pulpitis (SIP) assessed by CBCT followed by automated segmentation using Artificial intelligence (AI).

DETAILED DESCRIPTION:
Sixty human permanent molar teeth having irreversible pulpitis will be selected. Teeth will be randomly divided into 3 groups according to the type of pulpotomy; Group A: Photobiomodulation (PBM) pulpotomy, Group B: photocoagulation pulpotomy and Group C: Conventional pulpotomy which will serve as control. All 3 groups will be capped with bioceramic putty material. Post operative pain will be assessed at 24, 48 and 72 hours then after one week using numerical rating scale (NRS). Clinical and radiographic assessment using periapical radiograph of the healing progress will be done simultaneously during the follow up at one, three, six and 12 months intervals. CBCT will be done immediate postoperative and at the end of the follow up period to assess the dentin bridge formation and for automated segmentation to assess the radicular pulp volume changes.

ELIGIBILITY:
Inclusion Criteria:

* Permanent molar teeth with symptomatic irreversible pulpitis.
* The patient should be ≥ 16 to 50 years old.
* Teeth should give positive response to cold testing and clinical diagnosis of SIP with or without periapical rarefaction.
* Teeth will be selected only if they are restorable.
* Patient medically healthy and free from systemic diseases. ASA I, II.
* patients who agreed to participate in the study to attend the control visits.
* Teeth with periapical index score (PAI) 1 and 2 will be selected

Exclusion Criteria:

* Teeth with necrotic pulp, resorption or subgingival caries.
* Teeth with open apices.
* Medically compromised patients.
* Pregnant patients.
* Patients with uncontrollable bleeding from the radicular pulp.
* Patients with (PAI) score 3-5 will be excluded from the study

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of healing progress | one year
  evaluating clinically the signs and symptoms of pain and it will be recorded as yes and no question.
  -
Radiographic assessment of the dentin bridge formation | one year
  evaluating the dentin bridge formation using periapical radiographs and CBCT
Automated segmentation of the radicular pulp space | one year
  this will be done using CBCT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Rania Noaman ELbackly, Professor, Principal Investigator — Endodontics, Conservative Dentistry Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt. Tissue Engineering Laboratories, Faculty of Dentistry, Alexandria University, Alexandria, Egypt.
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No